CLINICAL TRIAL: NCT01408303
Title: A 6-Week, Randomized, Double-Blind, Placebo(Olive Oil)-Controlled Study to Assess the Efficacy and Safety of Add-On Epanova® to Statin Therapy in Subjects With Persistent Hypertriglyceridemia and High Risk for Cardiovascular Disease
Brief Title: [E]PANOVA Combined With a [S]TATIN in [P]ATIENTS With HYPERT[R]IGLYCER[I]DEMIA to Reduce Non-HDL CHOLES[T]EROL
Acronym: ESPRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Omthera Pharmaceuticals, Inc (Industry); Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OM-EPA-004; OM-EPA-004 (Other: Omthera Pharmaceuticals, Inc.); NCT01408303 (Other: ClinicalTrials.gov Identifier)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Hypertriglyceridemia; Cardiovascular Disease
Keywords: dyslipidemia; hyperlipidemia; cardiovascular risk
MeSH Terms: conditions — Hypertriglyceridemia; Cardiovascular Diseases; Dyslipidemias; Hyperlipidemias | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olive Oil (Placebo Comparator): olive oil: 4 g/day + prescription statin
  Interventions: Drug: Olive oil, 4g
- Epanova, 2 g (Experimental): omega-3-carboxylic acids, 2g/day + prescription statin
  Interventions: Drug: omega-3-carboxylic acids, 2g
- Epanova, 4 g (Experimental): omega-3-carboxylic acids, 4g/day + prescription statin
  Interventions: Drug: omega-3-carboxylic acids, 4g

INTERVENTIONS:
Drug: Olive oil, 4g — Olive oil: 4 x 1 g capsule daily for 6 weeks + prescription statin
  Other Names: Placebo comparator
  Arms: Olive Oil
Drug: omega-3-carboxylic acids, 2g — Epanova: 2 x 1 g capsule + olive oil 2 x 1 g capsule daily for 6 weeks + prescription statin
  Other Names: omega-3-carboxylic acids
  Arms: Epanova, 2 g
Drug: omega-3-carboxylic acids, 4g — Epanova: 4 x 1 g capsule daily for 6 weeks + prescription statin
  Other Names: omega-3-carboxylic acids
  Arms: Epanova, 4 g

SUMMARY:
The primary objective is to evaluate the efficacy of adding Epanova (2 g or 4 g daily) to an optimal statin monotherapy for lowering non-high-density lipoprotein (non-HDL) cholesterol in subjects with persistent hypertriglyceridemia and high risk for cardiovascular disease.

DETAILED DESCRIPTION:
The primary efficacy variable is serum non-HDL cholesterol. The primary endpoints are the differences in mean percent changes from baseline to end-of-treatment in non-HDL cholesterol between placebo and the 2g/day and 4g/day Epanova groups. Baseline is defined as the average of Visits 2, 3 and 4 (Weeks -2, -1 and 0) and end-of-treatment is the average of Visits 5 and 6 (Weeks 5 and 6).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, ≥18 years of age.
2. Fasting triglyceride (TG) level ≥200 mg/dL and <500 mg/dL.
3. The subject is a high risk for a future cardiovascular event.
4. The subject is treated with a statin and at or near LDL-C goal.

Exclusion Criteria:

1. Allergy or intolerance to omega-3 fatty acids and omega-3-acid ethyl esters.
2. Use of fibrates, bile acid sequestrants, or niacin or its analogues (greater than 200 mg/d) during screening.
3. Use of simvastatin 80 mg or Vytorin10/80 mg during screening.
4. Use of any eicosapentaenoic acid (EPA) or docosahexaenoic acid (DHA) products.
5. Use of any supplement for the purpose of lowering plasma cholesterol during screening.
6. Use of weight loss drugs or programs during screening.
7. Use of erythromycin, telithromycin, clarithromycin, cyclosporine, itraconazole, ketoconazole, protease inhibitors, or nefazodone during screening.
8. Use of anticoagulants during screening.
9. Use of oral or injected corticosteroids during screening.
10. Use of tamoxifen, estrogens, progestins, or testosterone, that has not been stable for >4 weeks at Visit 1, or is unstable during screening.
11. Use of >750 mL/d grapefruit juice during screening.
12. Known lipoprotein lipase impairment or deficiency, or apolipoprotein C-II deficiency or familial dysbetalipoproteinemia.
13. History of pancreatitis.
14. Type I diabetes mellitus, use of insulin, or HbA1c >10% at Visit 1.
15. Poorly controlled hypertension
16. Uncontrolled hypothyroidism, or thyroid stimulating hormone (TSH) >1.5xULN at Visit 2.
17. Recent history or current significant nephrotic syndrome, pulmonary, hepatic, biliary, gastrointestinal or immunologic disease.
18. History of cancer (except non-melanoma skin cancer, or carcinoma in situ of cervix) within the previous two years.
19. Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are not using an acceptable method of contraception.
20. Creatine kinase >5.0 times upper limit of normal (ULN); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times ULN at Visit 2.
21. Current or recent history (past 12 months) of drug or alcohol abuse.
22. Exposure to any investigational agent within 4 weeks prior to Visit 1.
23. Any other condition the investigator believes would interfere with the subject's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, MD, FACC, Study Director — Omthera Pharmaceuticals, Inc
Locations (81):
- United States (81):
  - Muscle Shoals, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Encinitas, California
  - Lomita, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Spring Valley, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Brandon, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Melbourne, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Oviedo, Florida
  - Ponte Vedra, Florida
  - St. Petersburg, Florida
  - Addison, Illinois
  - Chicago, Illinois
  - Oakbrook Terrace, Illinois
  - Indianapolis, Indiana
  - Newton, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Auburn, Maine
  - Oxon Hill, Maryland
  - Troy, Michigan
  - Edina, Minnesota
  - Chesterfield, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Endwell, New York
  - New Windsor, New York
  - Rochester, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Harleysville, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Rapid City, South Dakota
  - Bristol, Tennessee
  - Gray, Tennessee
  - Kingsport, Tennessee
  - Corpus Christi, Texas
  - Houston, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Olympia, Washington

REFERENCES:
- [Derived] Dunbar RL, Nicholls SJ, Maki KC, Roth EM, Orloff DG, Curcio D, Johnson J, Kling D, Davidson MH. Effects of omega-3 carboxylic acids on lipoprotein particles and other cardiovascular risk markers in high-risk statin-treated patients with residual hypertriglyceridemia: a randomized, controlled, double-blind trial. Lipids Health Dis. 2015 Sep 2;14:98. doi: 10.1186/s12944-015-0100-8. PMID 26328624
- [Derived] Maki KC, Orloff DG, Nicholls SJ, Dunbar RL, Roth EM, Curcio D, Johnson J, Kling D, Davidson MH. A highly bioavailable omega-3 free fatty acid formulation improves the cardiovascular risk profile in high-risk, statin-treated patients with residual hypertriglyceridemia (the ESPRIT trial). Clin Ther. 2013 Sep;35(9):1400-11.e1-3. doi: 10.1016/j.clinthera.2013.07.420. Epub 2013 Aug 30. PMID 23998969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period started August 2011 and the last subject visit was May 2012. All subjects were qualified at the clinical site and eligibility was determined by each PI (96 sites)
Pre-assignment Details: Subjects underwent 6-week washout and diet stabilization period, discontinued use of any non-statin lipid therapies, continued their current statin regimen, and followed the NCEP TLC diet. Men and women considered to be at high risk for atherosclerotic CVD and who had high serum TG (≥200 mg/dL and <500 mg/dL) were eligible for randomization.
Groups:
- Epanova, 2 g + Statin: omega-3 carboxylic acids, 1 g capsule
  omega-3 carboxylic acids + olive oil: omega-3 carboxylic acids 2 x 1 g capsule + olive oil 2 x 1 g capsule daily for 6 weeks
  prescribe statin
- Epanova, 4 g + Statin: omega-3 carboxylic acids, 1 g capsule
  omega-3 carboxylic acids: omega-3 carboxylic acids 4 x 1 g capsule daily for 6 weeks
  prescribed statin
- Olive Oil + Statin: olive oil, 1 g capsule
  olive oil: 4 x 1 g capsule daily for 6 weeks
  prescribed statin
Period: Overall Study
Arm/Group | Epanova, 2 g + Statin | Epanova, 4 g + Statin | Olive Oil + Statin
Started | 215 | 216 | 216
Completed | 209 | 204 | 210
Not Completed | 6 | 12 | 6
Not completed — Adverse Event | 3 | 7 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Noncompliance | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population comprised the Safety Population defined as subjects who received at least 1 dose of investigational product.
Groups:
- Epanova, 2 g: omega-3-carboxylic acids, 1 g capsule omega-3-carboxylic acids + placebo : omega-3-carboxylic acids 2 x 1 g capsule + placebo 2 x 1 g capsule daily for 6 weeks
- Epanova, 4 g: omega-3-carboxylic acids, 1 g capsule omega-3-carboxylic acids: omega-3-carboxylic acids 4 x 1 g capsule daily for 6 weeks
- Placebo: placebo, 1 g capsule
  placebo : 4 x 1 g capsule daily for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Epanova, 2 g | Epanova, 4 g | Placebo | Total
Number analyzed (Participants) | 215 | 216 | 215 | 646
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 138 | 141 | 124 | 403
  >=65 years | 77 | 75 | 91 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.95) | 60.1 (9.23) | 61.5 (9.64) | 60.8 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 79 | 93 | 264
  Male | 123 | 137 | 122 | 382
Region of Enrollment [Number; unit: participants]
  United States | 215 | 216 | 215 | 646

OUTCOME MEASURES:

1. Primary Outcome: Serum Non-HDL Cholesterol
Description: The primary endpoints are the differences in mean percent changes from baseline to end-of-treatment in non-HDL cholesterol between placebo and the 2g/day and 4g/day Epanova groups.
Time Frame: 6 weeks
Population: The Intent-to-Treat (ITT) Population was comprised of all subjects who were randomized. In the event that randomized subjects terminated before treatment or had no post-treatment efficacy assessments, a modified ITT Population was implemented."
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Groups:
- Epanova 2 g: omega-3-carboxylic acids, 1 g capsule omega-3-carboxylic acids + placebo: omega-3-carboxylic acids 2 x 1 g capsule + placebo 2 x 1 g capsule daily for 6 weeks
- Epanova 4 g: omega-3-carboxylic acids, 1 g capsule omega-3-carboxylic acids: omega-3-carboxylic acids 4 x 1 g capsule daily for 6 weeks
Arm/Group | Epanova 2 g | Epanova 4 g | Placebo
Number analyzed (Participants) | 209 | 207 | 211
Percent change from baseline | -3.86 [-7.316 to -0.277] | -6.91 [-10.204 to -3.504] | -0.91 [-4.509 to 2.822]
Statistical Analysis 1: Comparison: Epanova 2 g vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA; p-value from ANCOVA with factors for treatment, statin use and potency, and baseline value as a covariate, and adjusted using Hommel's procedure; LS mean difference relative to olive oil = -2.95
Statistical Analysis 2: Comparison: Epanova 4 g vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS mean difference relative to olive oil = -6.00

ADVERSE EVENTS:
Description: A total of 78 (12.1%) adverse events (AEs) were considered related to treatment: 13 in placebo, 21 in Epanova 2 g and 44 in Epanova 4 g. Twelve subjects (1.9%) had AEs causing discontinuation: 2 in placebo, 3 in Epanova 2 g and 7 in Epanova 4 g. Gastrointestinal disorders had the highest occurrence but most were mild or moderate and self-limiting.
Arm/Group | Epanova, 2 g | Epanova, 4 g | Placebo
Serious Adverse Events (participants affected / at risk) | 3/215 | 1/216 | 3/215
Other Adverse Events (participants affected / at risk) | 13/215 | 36/216 | 5/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova, 2 g (N=215) | Epanova, 4 g (N=216) | Placebo (N=215)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epanova, 2 g (N=215) | Epanova, 4 g (N=216) | Placebo (N=215)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 36 (36) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6) | 13 (13) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual investigators may publish data arising from their own subjects. The PI will provide the Sponsor with copies of written publications (including abstracts and posters)at least 60 days in advance of submission. Data will be reviewed by all participating investigators prior to publication. The Sponsor will have 60 days to review all definitive publications, such as manuscripts and book chapters, and a minimum of 30 days to review all abstracts.